CLINICAL TRIAL: NCT00477256
Title: Psychosocial Predictors of Child Adjustment and School Reintegration Outcome in a Pediatric Cancer Population
Brief Title: School Reintegration Outcomes in Pediatric Cancer Patients
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2007-0007
Record Dates: First submitted 2007-05-22; First posted 2007-05-23 (Estimated); Last update posted 2012-07-31 (Estimated); Status verified 2012-07

CONDITIONS: Pediatric Cancers
Keywords: Pediatric Cancer; Child Adjustment; School Reintegration; Caregiver; Questionnaire; Quality of Life; Survey
MeSH Terms: conditions — Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Child: Children between 6 and 17 years diagnosed with, and treated for, any type of cancer.
  Interventions: Behavioral: Questionnaires
- Parent: Parent(s) or caregiver(s) of children with cancer.
  Interventions: Behavioral: Questionnaires
- Medical Staff: Medical staff (i.e., physicians, nurse practitioners) involved in the children's medical decision-making.
  Interventions: Behavioral: Questionnaires

INTERVENTIONS:
Behavioral: Questionnaires — 5 Paper-and-Pencil Questionnaires: All participants will engage in a one-time completion of all measures.
  Other Names: Survey

SUMMARY:
Primary Objectives:

1. To examine illness-related factors (i.e., severity of illness, quality of life rating) as predictors or correlates of child adjustment to pediatric cancer.
2. To examine illness-related factors (i.e., severity of illness, quality of life rating) as predictors of school reintegration (i.e., school attendance) in children with pediatric cancer.
3. To examine a within-parent factor (i.e., parental stress) as a predictor or correlate of child adjustment to pediatric cancer.
4. To examine a within-parent factor (i.e., parental stress) as a predictor or correlate of school reintegration (i.e., school attendance).

Secondary Objectives:

1. To examine a second within-parent factor (i.e., parental perception of child vulnerability) as a predictor or correlate of child adjustment to pediatric cancer.
2. To examine a second within-parent factor (i.e., parental perception of child vulnerability) as a predictor or correlate of school reintegration (i.e., school attendance) in children with pediatric cancer.
3. To develop a statistical model by which relative contributions of each predictor variable (i.e., severity of illness, quality of life, parental stress, parental perception of child vulnerability), as well as their interrelatedness, can be understood in relation to child adjustment. Exploration of each variable's contribution will affect the schematic organization of the model.
4. To examine demographic variables as covariates in the primary analyses. The variables include: child's age, gender, grade, ethnicity, diagnosis, time since diagnosis, type and duration of treatment, and time since school reintegration.

DETAILED DESCRIPTION:
Consent for Child Participation:

STUDY PARTICIPATION:

If you agree to take part in this study, you will complete 3 paper-and-pencil questionnaires that will be used to get information about your health status and overall well being. You will be asked how you are feeling at this time, whether you worry a lot of the time, how often you feel sad, and how physically active you are, such as with walking and running. The study staff is also interested in knowing how well you are keeping up with school activities and how often you attend school. Finally, your doctor will provide information about your illness and describe how it may affect your participation at home or at school.

If you are age 8 or above, it should take about 30-45 minutes to complete the questionnaires. If you are between age 6 and 7, it should take about 10-15 minutes to complete the questionnaires.

Your parent or caregiver may be present while you complete your questionnaires. However, you are encouraged you to give your own answers. The questionnaires may be completed in The Children's Cancer Hospital clinic or elsewhere, and a research assistant will assist you, if you need help.

Length of Study:

Your participation in this study will be over once you have completed the 3 questionnaires.

This is an investigational study. Up to 106 children will take part in this study. All will be enrolled at M. D. Anderson.

Consent for Medical Staff Participants:

Child Adjustment to Pediatric Cancer and School Reintegration:

Researchers want to examine illness-related factors (such as severity of illness and quality of life) as predictors or correlates of adjustment to pediatric cancer and predictors of school reintegration (such as school attendance) of children with pediatric cancer.

Study Participation:

If you agree to take part in this study, you will complete one, 7-item paper-and-pencil measure that will be used to obtain information about your patient's current health status. For example, the first question asks, "On a Likert scale of 1 to 7, describe the degree of impairment for this child." One (1) indicates "Independent functioning, requires no assistance," and 7 indicates "Requires complete assistance." It should take about 2-5 minutes to complete the measure in the clinic or your office, and it can be done during regular work hours.

You will also be asked to describe information on the child's severity of illness. For example, you will be asked to describe the degree of impairment, frequency of medical procedures/hospitalizations, and your understanding of the child's participation in community activities.

Length of Study:

Your participation in this study will be over once you have completed the measure. Study results will be published and mailed to each medical staff participant.

This is an investigational study. Up to 24 medical staff members will take part in this study. All will be enrolled in this study at M. D. Anderson.

Consent for Parent or Caregiver Participation:

Child Adjustment to Pediatric Cancer and School Reintegration:

Researchers want to learn about illness-related factors (such as severity of illness and quality of life) that may show how well children with cancer adjust to the disease and return to a traditional school setting (by looking at school attendance, for example).

Your Study Participation:

If you agree to take part in this study, you will complete 5 paper-and-pencil questionnaires that will be used to get information about you and your child's health status. Questions will be about your child's physical, emotional, and social functioning as well as how they are functioning in school. You will be asked to rate how much of a problem you think your child may be having in these areas. You will also be asked about how often difficult events have occurred for you as a parent or caregiver of a child with cancer. These questionnaires should take about 45 minutes to 1 hour to complete.

The Child's Participation:

Your child will also be asked to complete 3 paper-and-pencil questionnaires that will also be used to get information about his or her health status, as well as his or her overall well being.

You may be present with your child while he or she is completing the questionnaires, if you choose. However, you are encouraged to allow the child to complete the questionnaires on his or her own so as not to influence the child's answers. A research assistant will be glad to assist your child with his or her completion of the questionnaires.

Location for Completion of Questionnaires:

The questionnaires for both you and the child may be completed in a private consultation room or examination room in The Children's Cancer Hospital clinic, or they may be completed outside of the room or clinic and returned to study staff.

If they are completed outside of the room or clinic, you can hand deliver the questionnaires to the clinic in an envelope, or you can mail them back to study staff in a postage-paid return envelope that can be provided to you.

Length of Study:

Your participation in this study will be over once you have completed the 5 questionnaires. You may receive a summary of the study's findings at the end of the study if you make this request to the study researcher who gave the questionnaires to the study doctor.

This is an investigational study. Up to 106 parents or caregivers will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Children between 6 and 17 years diagnosed with, and treated for, any type of cancer
2. Children enrolled in grades K through 12
3. Children who have actively participated in community or private school during the 2006-2007 academic year
4. Children who have experienced a period of absence from community or private school of at least two consecutive months as a result of medical treatment prior to school reintegration
5. Children who have fully reintegrated as a full-time student within the past 1-3 years
6. Parents and children who are either English- or Spanish-speaking and are able to read in either or both languages
7. Medical staff (i.e., physicians, nurse practitioners) involved in the children's medical decision-making

Exclusion Criteria:

1. Children and/or parents diagnosed and/or identified as having mental retardation (IQ < 70) with concomitant adaptive behavior deficits or classified as having any type of Pervasive Developmental Disorder (PDD)
2. Children and/or parents who speak a language other than English or Spanish
3. Participant (e.g., parent or child) unwillingness to participate in any capacity

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children between 6 and 17 years diagnosed with, and treated for, any type of cancer, their parent(s) or caregiver(s), and medical staff (i.e., physicians, nurse practitioners) involved in the children's medical decision-making.
Sampling Method: Probability Sample
Enrollment: 91 (Actual)
Dates: Start 2007-05; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Severity of Illness [using The Severity of Illness Scale (SOIS)] | Completion of scale by medical staff, approximately 2-5 minutes
Quality of Life [using The Pediatric Quality of Life (PedsQL)] | Questionnaire, approximately 45 minutes to one hour for parent or non-parent caregivers to complete their measures

CONTACTS AND LOCATIONS:
Overall Officials: Martha Askins, PhD, BA, MA, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center website — http://www.mdanderson.org